CLINICAL TRIAL: NCT03689062
Title: Premature Rupture of Membranes at 34 to 37 Weeks' Gestation :Active vs Conservative Management
Brief Title: Premature Rupture of Membranes at 34 to 37 Weeks' Gestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Abd El Sattar Ahmed, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROM
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Premature Rupture of Membrane
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Labor, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservative group (Active Comparator): patient assigned to the observation group will be assessed in the labor and delivery suite for 2 to 4 hours with continuous external fetal heart rate monitoring and tocodynamometry. In the absence of non reassuring fetal status , initiation of labor , or infection , these women will be transferred to antepartum room where maternal vital signs. Patients will be restricted to bed rest with bathroom privileges and remained hospitalized until delivary .
  Interventions: Procedure: follow up
- active group (Experimental): Patients assigned to active management will receive induction of labour with intravenous oxytocin with use of controlled infusion pump Oxytocin will be administered by continuous intravenous infusion beginning at 0.5 mU/min , doubling the dose every 30 minutes to 2mU/min , and then increasing by 2 mU/min every 30 minutes there after until a satisfactory labor pattern is achieved.
  Interventions: Procedure: induction of labor

INTERVENTIONS:
Procedure: induction of labor — oxytocin intravenous drip
  Arms: active group
Procedure: follow up — hospitalization and antibiotics
  Arms: conservative group

SUMMARY:
Prelabour rupture of membrane is deﬁned as rupture of membranes prior to the onset of labour. Approximately 8% of pregnant women at term experience PROM, but the decision as to how term PROM should be managed clinically remains controversial, and there is wide variation in practice with no clear consensus on what constitutes optimal treatment. Although for the majority of women labour will start spontaneously within 24 hours following term PROM, up to 4%of women will not experience spontaneous onset of labour within seven days.

ELIGIBILITY:
Inclusion Criteria:

* Preterm premature rupture of membranes.
* Singleton gestation.
* Pregnant between 34 weeks 0 days to 36 weeks 6 days.

Exclusion Criteria:

* Non cephalic presentation.
* fetal distress.
* Labour on admission.
* Medical or obstetric complications such as(suspected chorioamnionitis ,hypertensive disorders, diabetes mellitus , active genital herpes , placenta previa , infection, meconium stained amniotic fluid ,severe fetal anomalies).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients with chorioamnionitis | 24 hours
  Clinical chorioamnionitis is defined in the absence of other causes of hyperpyrexia by a temprature of >38 C with either uterine tenderness , leucocytosis , maternal or fetal tachycardia , or foul smelling vaginal discharge